CLINICAL TRIAL: NCT04446520
Title: Autogenic Drainage Effect on Blood Gases and Prevention of Pulmonary Complication After Upper Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Princess Nourah Bint Abdulrahman University (Other)
Responsible Party: Principal Investigator, Mona Mohamed Taha, ASSISTANT PROFESSOR, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P.T REC/012/001740
Record Dates: First submitted 2020-06-21; First posted 2020-06-25 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Postoperative Complications
Keywords: Autogenic drainage; blood gases; Pneumonia,; upper abdominal surgery; Postoperative pulmonary Complications
MeSH Terms: conditions — Postoperative Complications; Pneumonia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- autogenic drainage and traditional physiotherapy (Experimental): autogenic drainage technique plus traditional physiotherapy (localized breathing exercise, diaphragmatic breathing and splinted coughing)
  Interventions: Procedure: autogenic drainage
- traditional physiotherapy (Active Comparator): traditional physiotherapy (localized breathing exercise, diaphragmatic breathing, and splinted coughing)
  Interventions: Procedure: autogenic drainage

INTERVENTIONS:
Procedure: autogenic drainage — breathing control using expiratory airflow to mobilize secretions from smaller to larger airways. Secretions are cleared independently by adjusting the depth and speed of respiration in a sequence of controlled breathing techniques during exhalation in addition to traditional physiotherapy (deep breathing exercise, diaphragmatic breathing and splinted coughing)

SUMMARY:
Purpose: This study will find out the effect of Autogenic drainage on the prevention of pulmonary complications after upper abdominal surgery. Method: Sixty patients post upper abdominal surgeries will be included, their ages ranged from 50 to 60 years old. The patients will be divided into two groups, study group (A) include patients that receive first traditional physiotherapy (localized breathing exercise, diaphragmatic breathing, and splinted coughing) then autogenic drainage (B)-Group B: patients that receive traditional physiotherapy (localized breathing exercise, diaphragmatic breathing and splinted coughing)

DETAILED DESCRIPTION:
Purpose: This study will find out the effect of Autogenic drainage on the prevention of pulmonary complications after upper abdominal surgery. Method: Sixty patients post upper abdominal surgeries will be included, their ages ranged from 50 to 60 years old. The patients will be divided into two groups, study group (A) include patients that receive first traditional physiotherapy (localized breathing exercise, diaphragmatic breathing, and splinted coughing) then autogenic drainage (B)-Group B: patients that receive traditional physiotherapy (deep breathing exercise, diaphragmatic breathing and splinted coughing)

ELIGIBILITY:
Inclusion Criteria:

* Age from 50 to 60 years
* Patients undergoing elective upper abdominal surgery with an abdominal incision longer than 5 cm that is above or extending above the umbilicus.
* Non-smoker patients

Exclusion Criteria:

* Patients developing cancer
* Patients with rib fractures
* Inability to comprehend and follow instructions.
* Pre-existing obstructive sleep apnea
* Current hospital patient for a separate episode of care.
* Patients requiring esophageal surgery or organ transplant.

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-06-27 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-09-05 (Actual)

PRIMARY OUTCOMES:
arterial blood gases | 7 days

SECONDARY OUTCOMES:
prevalence of post operative pulmonary complication (pneumonia, hypoxemia and atelectasis) and number of days staying in ICU | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Mona Taha, PhD, Principal Investigator — Cairo University
Locations (1):
- Kasr Alaini, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Taha MM, Draz RS, Gamal MM, Ibrahim ZM. Adding autogenic drainage to chest physiotherapy after upper abdominal surgery: effect on blood gases and pulmonary complications prevention. Randomized controlled trial. Sao Paulo Med J. 2021 Nov 15;139(6):556-563. doi: 10.1590/1516-3180.2021.0048.0904221. eCollection 2021. PMID 34787294